CLINICAL TRIAL: NCT07040475
Title: Effects of the Clinical Application of TCIM Procedures During Inpatient Stays in Germany - a Multicenter Observational Study
Brief Title: Effects of the Clinical Application of Traditional, Complementary and Integrative Medicine (TCIM) Procedures During Inpatient Stays in Germany
Acronym: Minerva
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Universität Tübingen (Other); Universität Duisburg-Essen (Other); Sozialstiftung Bamberg (Other)
Responsible Party: Principal Investigator, Michael Jeitler, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: Minerva
Record Dates: First submitted 2025-06-11; First posted 2025-06-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TCIM
  Interventions: Other: Inpatient TCIM therapy

INTERVENTIONS:
Other: Inpatient TCIM therapy — This multicenter, prospective, uncontrolled observational study is evaluating the effects and safety of inpatient TCIM therapy (German: naturheilkundliche Komplextherapie) at three German clinics: Immanuel Hospital Berlin, Klinikum Bamberg, and Evangelical Clinics Essen-Mitte. This therapy, reimbursed by statutory health insurance under certain conditions, combines evidence-informed TCIM approaches such as hyperthermia, exercise therapy, phytotherapy, and dietary interventions including fasting i.a.

SUMMARY:
The aim of this healthcare research project is to evaluate the effects of routine inpatient TCIM (Traditional, Complementary and Integrative Medicine) care in Germany. The focus is on the TCIM centers at Immanuel Krankenhaus Berlin, Klinikum Bamberg und Evang. Kliniken Essen-Mitte, where inpatient TCIM therapies are to be systematically evaluated. This form of therapy, which is reimbursed by statutory health insurance providers (under certain conditions), is based on a combination of various evidence-based TCIM approaches. These include hyperthermia, exercise therapy, Mind-Body Medicine, phytotherapy, nutritional therapy, fasting therapy inter alia.

ELIGIBILITY:
Inclusion criteria:

* Beginning (first 24 hours) inpatient TCIM treatment at Immanuel Hospital Berlin, Bamberg Hospital, or Evangelische Kliniken Essen-Mitte
* Written consent form

Exclusion criteria:

* Insufficient language skills
* Dementia or other severely impairing cognitive disorders
* Pregnancy or breastfeeding
* Participation in a clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in TCIM wards are offered the opportunity to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Form Health Survey - 12 Items (SF-12) | Baseline, 3 months
  0-100, higher scores indicate better health status.

SECONDARY OUTCOMES:
Short Form Health Survey - 12 Items (SF-12) | Baseline, up to 14 days, 6 months, 12 months
  0-100, higher scores indicate better health status.
EuroQol 5-Dimension 5-Level | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0 (worst) to 1 (best), higher scores indicate better health-related quality of life.
Food Frequency List | Baseline, up to 14 days, 3 months, 6 months, 12 months
  Descriptive measure; not scored on a numeric scale.
International Physical Activity Questionnaire - Short Form | Baseline, up to 14 days, 3 months, 6 months, 12 months
  MET-min/week (variable), higher scores indicate higher physical activity levels.
Hospital Anxiety and Depression Scale | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-21 per subscale (Anxiety and Depression), higher scores indicate more severe symptoms.
Work Productivity and Activity Impairment Questionnaire | Baseline, 3 months, 6 months, 12 months
  0%-100%, higher scores indicate greater impairment (i.e., worse outcome).
Perceived Stress Scale - 4 | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-16, higher scores indicate higher perceived stress.
Main complaint | Baseline, up to 14 days, 3 months, 6 months, 12 months
  Visual Analog Scale (0-100, higher scores mean a worse outcome)
Fibromyalgia Impact Questionnaire | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-100, higher scores indicate greater impact of fibromyalgia (worse outcome).
Rheumatoid Arthritis Disease Activity Index | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-10, higher scores indicate greater disease activity (worse outcome).
Bath Ankylosing Spondylitis Disease Activity Index | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-10, higher scores indicate more active disease (worse outcome).
Bath Ankylosing Spondylitis Functional Index | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-10, higher scores indicate more functional limitation (worse outcome).
Western Ontario and McMaster Universities Osteoarthritis Index | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-100, higher scores indicate greater pain/stiffness/disability (worse outcome).
Irritable Bowel Syndrome Symptom Severity Score | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-500, higher scores indicate more severe IBS symptoms (worse outcome).
Short Inflammatory Bowel Disease Questionnaire | Baseline, up to 14 days, 3 months, 6 months, 12 months
  10-70, higher scores indicate better quality of life.
Pain Disability Index | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-70, higher scores indicate greater disability (worse outcome).
Roland Morris Disability Questionnaire | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-24, higher scores indicate more severe disability (worse outcome).
Maslach Burnout Inventory | Baseline, up to 14 days, 3 months, 6 months, 12 months
  Variable by subscale (Emotional Exhaustion: 0-54, Depersonalization: 0-30, Personal Accomplishment: 0-48) Higher scores on EE/DP = worse outcome; higher PA = better outcome.
Beck Depression Inventory-II | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-63, higher scores indicate more severe depressive symptoms (worse outcome).
Diabetes Distress Scale - 2 | Baseline, up to 14 days, 3 months, 6 months, 12 months
  1-6, higher scores indicate greater emotional distress related to diabetes (worse outcome).
Dermatology Life Quality Index | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-30, higher scores indicate greater impact on quality of life (worse outcome).
Functional Assessment of Cancer Therapy - General | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-108, higher scores indicate better quality of life.
Use of the healthcare system | Baseline,12 months
  Descriptive data (e.g., number of visits); not a scored scale.
Expectations regarding inpatient TCIM treatment | Baseline
  5-point Likert scale, 1-5. Higher scores indicate stronger or more positive expectations.
Chalder Fatigue Scale | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-33, higher scores mean a worse outcome
Somatic Symptom Scale | Baseline, up to 14 days, 3 months, 6 months, 12 months
  0-32, higher scores mean a worse outcome
Body weight [kg] | Baseline, up to 14 days
Height [in cm] | Baseline
BMI [kg/m2] | Baseline, up to 14 days
Systolic blood pressure [mmHg], diastolic blood pressure [mmHg] | Baseline, up to 14 days
Waist circumference [in cm] | Baseline, up to 14 days
Triglycerides [mg/dl] | Baseline, up to 14 days
Total cholesterol [mg/dl] | Baseline, up to 14 days
HDL [mg/dl] | Baseline, up to 14 days
LDL [mg/dl] | Baseline, up to 14 days
Glucose [mg/dl] | Baseline, up to 14 days
Uric acid [μmol/L] | Baseline, up to 14 days
Creatinine [mg/dl] | Baseline, up to 14 days
CRP [mg/l] | Baseline, up to 14 days
GPT [U/l] | Baseline, up to 14 days
HbA1c [mmol/mol] | Baseline, up to 14 days
HbA1c [%] | Baseline, up to 14 days
Headache Impact Test (HIT-6) | Baseline, up to 14 days, 3 months, 6 months, 12 months
  36-78. A higher value indicates a greater impairment due to headaches.
Integrity of the duodenal intestinal barrier analyzed by confocal laser endomicroscopy (CLE) | Baseline, within 3 to 12 months
  The integrity of the intestinal barrier is tested via CLE during routine esophagogastro-duodenoscopy to detect primary or secondary (food-induced) barrier defects.
  By CLE, the intestinal mucosa and the epithelial lining can be analyzed in vivo with a 1000 x magnification. An intestinal barrier defect can be detected by the leakage of a contrast agent (fluorescein) from the blood vessels through the intestinal epithelial spaces into the intestinal cavity and the shedding of epithelial cells.
Result of the esophagogastro-duodenoscopy | Baseline, within 3 to 12 months
  Participants undergo an esophagogastro- duodenoscopy with CLE when clinically indicated as part of their inpatient care. Thereby, the inflammatory status and the intestinal barrier is routinely analyzed.
Histopathological analysis of duodenal biopsies | Baseline, within 3 to 12 months
  Intestinal biopsies, which are routinely taken during esophagogastroduodenoscopy, are processed for histopathological analysis of the mucosal and epithelial structure as well as of the immune cell compartment and to rule out inflammatory processes or intestinal infections.
Immunohistochemical analysis of duodenal biopsies | Baseline, within 3 to 12 months
  Intestinal biopsies, which are routinely taken during esophagogastroduodenoscopy, are stained using immunohistochemistry and examined for the expression of specific marker proteins (e.g. CD3, eosinophils, Occludin, Claudins).
IgE antibody titers | Baseline, within 3 to 12 months
  IgE screening of antibodies against typical food allergens (egg white, soy, milk, yeast, wheat) in the serum
Analysis of fecal biomarkers, digestive parameters, intestinal flora | Baseline, within 3 to 12 months
  The concentrations of different fecal biomarkers are analyzed in stool samples:
  Calprotectin, Lactoferrin, PMN-Elastase, EDN, Zonulin, Alpha-1-Antitrypsin, Beta-Defensin.
  Furthermore, digestive parameters such as digestion residues and the intestinal flora are determined.
Result of hydrogen breath tests | Baseline, within 3 to 12 months
  Lactose, fructose, and sorbitol intolerance is tested via hydrogen breath test

OTHER OUTCOMES:
Number of participants with diagnoses | Baseline, up to 14 days, 3 months, 6 months, 12 months
Number of participants taking pain medication | Baseline, up to 14 days, 3 months, 6 months, 12 months
Number of participants taking antidepressive medication | Baseline, up to 14 days, 3 months, 6 months, 12 months
Number of participants taking anxiolytics | Baseline, up to 14 days, 3 months, 6 months, 12 months
Number of participants taking migraine medication | Baseline, up to 14 days, 3 months, 6 months, 12 months
Number of participants taking antihypertensive medication | Baseline, up to 14 days, 3 months, 6 months, 12 months
Number of participants taking lipid-lowering medication | Baseline, up to 14 days, 3 months, 6 months, 12 months
Number of participants taking corticosteroids | Baseline, up to 14 days, 3 months, 6 months, 12 months
Number of participants taking antidiabetic medication | Baseline, up to 14 days, 3 months, 6 months, 12 months
Number of participants taking biologics | Baseline, up to 14 days, 3 months, 6 months, 12 months
Number of participants taking immunosuppressants | Baseline, up to 14 days, 3 months, 6 months, 12 months
Adverse events | Baseline, up to 14 days, 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Sozialstiftung Bamberg, Klinikum Bamberg, Bamberg
  - Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Institut für Sozialmedizin, Epidemiologie und Gesundheitsökonomie, Charité - Universitätsmedizin Berlin, Berlin
  - Klinik für Naturheilkunde und Integrative Medizin, KEM, Essen